CLINICAL TRIAL: NCT00963846
Title: Huperzine for Cognitive and Functional Impairment in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedisyn Corporation (Industry)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Scott Woods, MD, Consultant, Biomedisyn Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Biomedisyn 200901; 3R41MH083436-01A1S1 (NIH)
Record Dates: First submitted 2009-08-10; First posted 2009-08-24 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognition; functioning
MeSH Terms: conditions — Schizophrenia | interventions — huperzine A; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- huperzine 0.2 mg BID (Experimental)
  Interventions: Drug: huperzine 0.2 mg BID
- huperzine 0.4 mg BID (Experimental)
  Interventions: Drug: huperzine 0.4 mg BID
- huperzine 0.8 mg BID (Experimental)
  Interventions: Drug: huperzine 0.8 mg BID

INTERVENTIONS:
Drug: placebo — matching pill placebo
  Arms: placebo
Drug: huperzine 0.2 mg BID — huperzine rising doses up to 0.2 mg BID
  Arms: huperzine 0.2 mg BID
Drug: huperzine 0.4 mg BID — huperzine rising doses up to 0.4 mg BID
  Arms: huperzine 0.4 mg BID
Drug: huperzine 0.8 mg BID — huperzine rising doses up to 0.8 mg BID
  Arms: huperzine 0.8 mg BID

SUMMARY:
Huperzine is a natural plant product with procognitive properties in patients with Alzheimer's disease. Cognitive difficulties hamper functioning in schizophrenia as well. The present study will investigate whether huperzine improves cognition and functioning in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Psychiatric diagnosis of schizophrenia according to SCID-IV.
2. Currently treated with an antipsychotic medication.
3. Has tolerated current antipsychotic treatment adequately.
4. Has received an adequate trial of antipsychotic (a least 3 months of at least 300 mg/d CPZ equivalent).
5. Has been receiving current psychotropic medication (s) for at least 8 weeks.
6. Has been receiving current doses of psychotropic medication (s) for at least 4 weeks.
7. Has been clinically stable for at least 12 weeks.
8. No more than moderate severity (4 on the 1-7 scale) on any PANSS positive item.
9. No more than 15 on the total of PANSS negative symptom items.
10. Simpson-Angus Scale total score <7.
11. Calgary Depression Scale for Schizophrenia total score <11.
12. Submaximal performance on at least one of the following MATRICS components (letter-number span <20 OR HVLT total <31 OR CPT d-prime < 3.47).
13. Score > 1 SD below age-, gender-, and education-adjusted normal control mean on MATRICS composite
14. Good general health with no additional diseases expected to interfere with the studies.
15. Fluent in English.
16. Age 18-55.
17. Adequate visual and auditory acuity to allow neuropsychological testing.
18. Able to ingest oral medication.
19. Not pregnant or lactating (women of childbearing potential must use a medically accepted method of birth control).
20. Onset of schizophrenia prior to age 45.
21. Available informant knowledgeable about subject's current functioning.
22. Informed consent obtained from the subject prior to entry into the study.

Exclusion Criteria:

1. Poor reading skills (raw score on MATRICS Wechsler Test of Adult Reading < 6).
2. History of systemic cancer within 5 years.
3. Use of any investigational drugs within 30 days prior to the screening visit.
4. Use of cholinesterase inhibitors (galantamine, rivastigmine, donepezil, or tacrine) within 4 weeks of screening.
5. Any clinically significant laboratory test abnormality on screening tests (hematology, chemistry, urinalysis, EKG). Clinically significant LFT elevations will be defined as >2x the upper limit of normal.
6. Any significant neurologic disease including Alzheimer's disease, parkinson's disease, stroke, huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, history of head injury with loss of consciousness for greater than one day within the past 5 years, or with residual deficits.
7. Use of antihypertensive agents with frequent CNS side effects (e.g. clonidine, propranolol) within 4 weeks prior to the screening visit.
8. Use of medications known to alter drug absorption or metabolism (e.g. probenecid, cimetidine, anti-fungal agents, erythromycin, rifampin, and anticonvulsants) within 4 weeks prior to the screening visit.
9. History of peptic ulcer disease within 2 years.
10. History of myocardial infarction, significant cardiovascular disease, or congestive heart failure within 6 months, history of hepatic or renal insufficiency, insulin-requiring diabetes or uncontrolled diabetes mellitus.
11. Clinically significant cardiac arrhythmia, resting pulse less than 50.
12. Present use or use in the 4 weeks prior to screening of anti-parkinsonian or anticholinergic medications (e.g. Sinemet, amantadine, bromocriptine, pergolide, selegiline, atropine, scopolamine, benztropine, trihexyphenidyl, hydroxyzine, diphenhydramine).
13. Use of narcotic analgesics within 4 weeks prior to the screening visit.
14. History of alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria).
15. Receiving CYP 1A2 inhibitors such as certain SSRIs (all excluded in #4) cimetidine, methoxsalen, quinolones, furafylline, or moclobemide.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
MATRICS battery | 26 weeks

SECONDARY OUTCOMES:
UPSA | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Biomedisyn Corporation
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States